CLINICAL TRIAL: NCT02679014
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose, Parallel Study to Investigate the Pharmacokinetics, Pharmacodynamic Effects, Safety and Tolerability of Repeated Dosing of RO5459072 in Volunteers With Celiac Disease
Brief Title: A Study to Investigate the Pharmacokinetics, Pharmacodynamic Effects, Safety and Tolerability of Repeated Dosing of RO5459072 in Volunteers With Celiac Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP29911; 2015-002864-18 (EudraCT Number)
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — petesicatib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo capsules (2 capsules) twice daily for 28 days.
  Interventions: Drug: Placebo
- RO5459072 (Experimental): Participants will receive RO5459072 100 milligrams (mg) capsules (2*50 mg capsules) twice daily for 28 days.
  Interventions: Drug: RO5459072

INTERVENTIONS:
Drug: Placebo — With the exception of the mornings of Days 7 and 21, placebo capsules will be taken orally with a glass of still water in the morning and evening under fed conditions. On the mornings of Days 7 and 21, placebo will be administered under fasted conditions (overnight fast of at least 8 hours before dosing).
  Arms: Placebo
Drug: RO5459072 — With the exception of the mornings of Days 7 and 21, RO5459072 capsules will be taken orally with a glass of still water in the morning and evening under fed conditions. On the mornings of Days 7 and 21, RO5459072 will be administered under fasted conditions (overnight fast of at least 8 hours before dosing).
  Other Names: RG7625
  Arms: RO5459072

SUMMARY:
A randomized, double-blind, placebo-controlled, two treatment, parallel group study to investigate the effects of RO5459072, a cathepsin S inhibitor, on the immune response to a gluten challenge in volunteers with celiac disease. Volunteers with previously diagnosed celiac disease will be randomized to receive either 100 milligrams (mg) RO5459072 or placebo twice daily with food for 28 days (Days 1 to 28).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with a biopsy confirmed diagnosis of celiac disease
* Human leukocyte antigen (HLA) serotype DQ 2.5 and HLA-DQ 8 haplotypes
* Maintaining a gluten-free diet for at least one year. Compliance will be assessed by serology, compatible responses to a self-reported assessment of gluten-free diet adherence and the absence of typical celiac disease symptoms
* Able to participate and to comply with the study restrictions including the requirements of the gluten challenge

Exclusion Criteria:

* A diagnosis of non-celiac gluten sensitivity
* A personal history of food intolerance other than to gluten, or diagnosis of galactosemia, lactose, galactose or fructose intolerance
* A personal history of severe acute symptomatic reaction to sporadic gluten ingestion
* A diagnosis of refractory celiac disease or presence of severe complications of celiac disease
* Diagnosed or suspected immunoglobulin A (IgA) deficiency
* Acute inflammatory bowel disease (ulcerative colitis, Crohn's disease), gastrointestinal obstruction or sub-occlusive syndromes, digestive perforation or risk of digestive perforation, painful abdominal syndromes of undetermined cause
* A history of stomach or intestinal surgery or resection. Appendectomy and hernia repair are acceptable
* Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple allergies (non-active hay fever is acceptable)
* Immunocompromised or with reduced immune function considered to be clinically significant by the Investigator
* Immunization within 30 days before the screening visit or planning vaccination during the study
* Women who are pregnant or lactating, or who are of child-bearing potential and do not agree to comply with requirements for contraceptive use. Men who do not agree to comply with requirements for contraceptive use and restrictions on sperm donation
* Participation in an investigational drug or device study within the three months preceding the screening visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-06 (Actual); Primary Completion 2016-08-28 (Actual); Study Completion 2016-08-28 (Actual)

PRIMARY OUTCOMES:
Overall Numbers of Participants who are Responders to the Gluten Challenge, Defined as Participants with an Increase in Number of Gliadin Specific T-cells Above Assay-Specific Thresholds | Day 13 and Day 29

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to Day 35
Number of Participants with an Increase in Antibody Titers (Anti-Tissue Transglutaminase [anti-tTG] Immunoglobulin A [IgA] and Immunoglobulin G [IgG] and Anti-Deamidated Gliadin Peptide (anti-DPG) IgA), as Determined Using Enzyme Immunoassay Methods | Screening, Day 7, Day 13, Day 21, Day 29 and Day 35 (Follow up)
Lactulose to Mannitol Ratio (LMR), Determined by Urine Concentrations of Lactulose and Mannitol | Day 7: 1 hour (hr) pre-dose to 1 hr post-dose, 1 hr to 3 hr post-dose, 3 hr to 5 hr post-dose and Day 21: 1 hr pre-dose to 1 hr post-dose, 1 to 3 hr post-dose, 3 hr to 5 hr post-dose
Change from Baseline in Number of Circulating White Blood Cells | Day 1 (Baseline), Day 7, Day 13, Day 21, and Day 29
Change from Baseline in Concentrations of the 10 kilodalton (kDa) Cluster of Differentiation 74 (CD74) Intermediate (Fragment p10) in B Cells | Day 1: pre-dose (=Baseline [BL]) and 4 hours (h) post-dose, Day 7: pre-dose and 4 h post-dose, Day 21: pre-dose and 4 h post-dose
Change from Baseline in Concentrations of Cathepsin S Mass Biomarker | Day 1 (Baseline), Day 7, Day 13, Day 21 and Day 29
Change from Baseline in Concentrations of Cystatin C Biomarker | Day 1 (Baseline), Day 7, Day 13, Day 21 and Day 29
Maximum Response (Emax ) in p10 upon Cathepsin S Inhibition Ex vivo | Day 1: pre-dose
Concentration of RO5459072 that Gives Half-maximal Response (EC50) in Ex Vivo p10 Stimulation Assay | Day 1: pre-dose
Change from Baseline in 4Beta-hydrocholesterol Concentration | Day 1 (Baseline), Day 7, Day 13, Day 21 and Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Hammersmith Medicines Research Ltd., London, United Kingdom

REFERENCES:
- [Derived] Bentley D, Mannino M, Manchester M, Teixeira PC, Reis B, Boyce M, Nagel S. A randomized, double-blind, placebo-controlled, multiple dose, parallel study to investigate the effects of a cathepsin S inhibitor in celiac disease. Clin Transl Sci. 2025 Jan;18(1):e13901. doi: 10.1111/cts.13901. PMID 39739628